CLINICAL TRIAL: NCT05165277
Title: Effect of Flow Rate and PH on Muscle Acidosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: TFDA terminated this study.
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Jiann-Her,Lin, Principal Investigator, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: N201909038
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Muscle Acidosis
Keywords: sngception; soreness; muscle acidosis; flow rate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acidic phosphate buffer solution (Experimental): The pH5.2 PBS will be given into the midpoint of the left tibialis muscle with flow rate of 0-40ml/hr for 2-26 minutes, that is, totally 5.5 ml of PBS.
  Interventions: Drug: Phosphate Buffer Solution
- Neutral phosphate buffer solution (Placebo Comparator): The pH 7.4 PBS will be given into the midpoint of the left tibialis muscle with flow rate of 0-40ml/hr for 2-26 minutes, that is, totally 5.5 ml of PBS.
  Interventions: Drug: Phosphate Buffer Solution

INTERVENTIONS:
Drug: Phosphate Buffer Solution — Phosphate-buffered saline (abbreviated PBS) is a buffer solution commonly used in biological research. It is a water-based salt solution containing disodium hydrogen phosphate, sodium dihydrogen phosphate. The buffer helps to maintain a constant pH. The osmolarity and ion concentrations of the solutions match those of the human body (isotonic).
  Other Names: Sodium phosphate solution; Phosphate buffered saline

SUMMARY:
This proposed study suggests that peripheral tissue acidosis sensed by the somatosensory system (sngception) would evoke the sng perception in the brain. This hypothesis is based on investigators preliminary data that the peripheral muscle acidosis will evoked the central sng perception. In this study, investigators want to determine if there is the correlation between the flow rate of drug application and sng or pain. Also, they try to find if the pH of a solution will affect muscle acidosis.

DETAILED DESCRIPTION:
Sng is a prominent complaint in Taiwanese people with low back pain. "Sng" is created to represent this Taiwanese word- 痠. Based on our preliminary data, sng was one of the most common complaints in patients with chronic low back pain (CLBP) and also one of the most common indication for lumbar spine operations. Back sng is not adequately relieved by pain-killers or even by the lumbar spine operations. By using functional MRI and questionnaires, our preliminary study demonstrated that sng is different from pain in the level of brain perception and the level of subjective concept. It is very likely that sng has its own unique nerve pathway other than pain. The subjective feeling of sng is very similar to sour in taste, so it is likely that acidosis may be involved in the process of sng sensation, especially in the muscle. Delayed onset muscle soreness is a well-known example, and the soreness is dependent on the proton-sensing neurons. Indeed, substantial evidences showed that up to 80% muscle afferents are acid-sensitive but not nociceptors. Therefore, the investigators propose that sng is the perception in the brain when the tissue acidosis is sensed by the somatosensory system, and "sng-ception" is created to indicate the sensation of tissue acidosis. However, the causal connection between the peripheral sngception and the central brain perception of sng is not established. The objective of this proposal is to establish the causal connection between peripheral muscle acidosis and the central brain sng perception. My central hypothesis is that acidosis-evoked sensation in the muscles will cause a central sng perception in the brain. This hypothesis is based on our previous studies that showed sng is different from pain in terms of subjective responses, brain activation areas and clinical impacts. To achieve this goal, two specific aims will be pursued 1. to determine if an acid solution will evokes sng response, and, 2.determining the correlation between the rate of drug application and muscle Sng. Successful establishment of the casual connection between the peripheral muscle acidosis and the central brain sng perception will lead to a more comprehensive understanding of sng mechanism and the potential medication development.

ELIGIBILITY:
Inclusion Criteria:

1. The subject ages ranges from 20-45 years old.
2. The subject has no chronic pain symptoms or complaint in last 6 months.
3. The subject is subjectively able to discriminate sng and pain.
4. The subject has no history of major diseases that required treatment or currently being under treatment.
5. Gender: men and women half
6. The used hand of subject is the right hand.
7. The educational level of subject is more than 9 years (graduated from junior high school)
8. The subject didn't have physical and mental illness
9. The subject didn't take prescribed medicine.
10. The VAS questionnaire must be 0 point both of low back "pain" and low back "soreness" assessment.
11. The subject who can fill the informed consent after understanding the purpose and medical help of this trial.

Exclusion Criteria:

1. The subject has:Neuropathic pain due to causes other than that specified in the inclusion criteria (e.g., post-herpetic neuralgia; painful diabetic neuropathy; mononeuritis multiplex; central poststroke pain; failed back surgery in relation to the presenting episode of radiculopathy; spinal abscess, infection, hematoma, or malignancy; phantom limb pain; peripheral neuropathy due to alcoholism, malignancy, human immunodeficiency virus [HIV], syphilis; drug abuse; vitamin B12 deficiency; hypothyroidism; liver disease; toxic exposure).

   Pain that is associated with a substantial somatic pain component (e.g., non-neuropathic/musculoskeletal pain in lower limbs or other parts of the body apart from the back) or more than one cause or potential cause for pain symptoms.Any painful concurrent rheumatic disease such as, but not limited to, fibromyalgia, rheumatoid arthritis, or significant osteoarthritis.
2. The subject is unable to reliably delineate or assess his or her own pain by anatomical location/distribution (e.g., the subject cannot reliably tell the difference between his or her back pain and lower limb pain and cannot rate the intensity of each separately).
3. The subject has undergone lumbar spine surgery within the last 6 months or has received treatment with epidural injections, nerve blocks, or acupuncture for LSR within 4 weeks before screening.
4. The subject had a malignancy according to his/her report.
5. The subject has had a positive test for HIV antibody or a history of HIV according to his/her report.
6. The subject has had a positive test for hepatitis B surface antigen or hepatitis C antibody according to his/her report.
7. The subject has a history of alcohol or narcotic substance abuse according to his/her report.
8. The subject is female and is pregnant or breastfeeding at the time of the screening visit or plans to become pregnant during the study period.
9. The subject cannot perform brain MRI scanning who had metal implants of head (such as fixed dentures, metal bone plate, vascular clamp, vascular embolization treatment coil, deep brain stimulator, artificial electronic ear, etc.), implants of head which affecting the image quality (such as the ventricle peritoneal catheter, etc.), implantation of permanent heart rate regulator, etc.
10. The subject has a history of spinal surgery.
11. The VAS questionnaire not be 0 point either low back "pain" or low back "soreness" assessment.
12. The subject has suffered from claustrophobia.
13. The subject has suffered from brain disease and had brain surgery.
14. The subject has taken prescribed medicine which can affect specific function of brian (such as sleeping pills, tranquilizer, etc.).
15. The subject has mental comorbidity (such as depression, panic disorder, etc)
16. The subject has mental retardation.
17. The educational level of subject is less than 9 years.
18. The subject ,who is unable to understand the purpose of this trial and fill the informed consent.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
The visual analog scale (VAS) of "sng" in the legs | Through completion of injection an average of 6 month
  The subject will be asked for sng VAS before infusion and immediately after infusion.
  Scale range 0 to 10 (1)0: No Sng (2)1-3: Mild Sng (3)4-6: Moderate Sng (4)7-9: Severe Sng (5)10: Worst Sng imaginable
The visual analog scale (VAS) of "pain" in the legs | Through completion of injection an average of 6 month
  The subject will be asked for pain VAS before infusion and immediately after infusion.
  Scale range 0 to 10 (1)0: No Pain (2)1-3: Mild Pain (3)4-6: Moderate Pain (4)7-9: Severe Pain (5)10: Worst Pain imaginable

SECONDARY OUTCOMES:
Muscle pressure pain threshold | Through completion of injection an average of 1 week
  Muscle pressure pain threshold on bilateral tibialis anterior muscles will be measured by algometer.

OTHER OUTCOMES:
36-Item Short Form Health Survey (RAND) | Up to 6 months before signing the informed consent form
  Investigator will evaluate the subject life quality and activity of daily life by 36-Item Short Form Health Survey (RAND) Consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Oswestry disability index | Up to 6 months before signing the informed consent form
  Investigator will evaluate the subject activity of daily life by Oswestry disability index The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100) (1)0 -20: Minimal disability (2)21-40: Moderate Disability (3)41-60: Severe Disability (4)61-80: Crippling back pain (5)81-100: These patients are either bed-bound or have an exaggeration of their symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Issberner U, Reeh PW, Steen KH. Pain due to tissue acidosis: a mechanism for inflammatory and ischemic myalgia? Neurosci Lett. 1996 Apr 26;208(3):191-4. doi: 10.1016/0304-3940(96)12576-3. PMID 8733302
- [Background] Law LAF, Sluka KA, McMullen T, Lee J, Arendt-Nielsen L, Graven-Nielsen T. Acidic buffer induced muscle pain evokes referred pain and mechanical hyperalgesia in humans. Pain. 2008 Nov 30;140(2):254-264. doi: 10.1016/j.pain.2008.08.014. Epub 2008 Oct 2. PMID 18835099
- [Background] Lin JH, Hung CH, Han DS, Chen ST, Lee CH, Sun WZ, Chen CC. Sensing acidosis: nociception or sngception? J Biomed Sci. 2018 Nov 29;25(1):85. doi: 10.1186/s12929-018-0486-5. PMID 30486810
- [Background] Fujii Y, Ozaki N, Taguchi T, Mizumura K, Furukawa K, Sugiura Y. TRP channels and ASICs mediate mechanical hyperalgesia in models of inflammatory muscle pain and delayed onset muscle soreness. Pain. 2008 Nov 30;140(2):292-304. doi: 10.1016/j.pain.2008.08.013. Epub 2008 Oct 1. PMID 18834667
- [Background] Chen CC, Wong CW. Neurosensory mechanotransduction through acid-sensing ion channels. J Cell Mol Med. 2013 Mar;17(3):337-49. doi: 10.1111/jcmm.12025. Epub 2013 Mar 14. PMID 23490035
- [Background] Chen WN, Lee CH, Lin SH, Wong CW, Sun WH, Wood JN, Chen CC. Roles of ASIC3, TRPV1, and NaV1.8 in the transition from acute to chronic pain in a mouse model of fibromyalgia. Mol Pain. 2014 Jun 23;10:40. doi: 10.1186/1744-8069-10-40. PMID 24957987